CLINICAL TRIAL: NCT06406543
Title: Vitamin D in Armenia: Phase 2 - Vitamin D Repletion Strategies With Dibase, and Vitamin D and Vitamin D Binding Protein and COVID
Brief Title: Vitamin D in Armenia: Vitamin D Repletion Strategies With Dibase, and Vitamin D and Vitamin D Binding Protein and COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Osteoporosis Center of Armenia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAT5256
Record Dates: First submitted 2024-05-07; First posted 2024-05-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D repletion
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose, high frequency vitamin D repletion (Experimental): receive 7,000 IU oral drops daily for 12 weeks, followed by 3,500 IU daily for 24 weeks
  Interventions: Dietary Supplement: Vitamin D3 (Cholecalciferol)
- Medium dose, medial frequency vitamin D repletion (Experimental): 50,000 IU oral solution weekly for 12 weeks, followed by 25,000 weekly for 24 weeks
  Interventions: Dietary Supplement: Vitamin D3 (Cholecalciferol)
- High dose, low frequency vitamin D repletion (Experimental): 100,000 IU every other week for 12 weeks, followed by 50,000 every other week for 24 weeks
  Interventions: Dietary Supplement: Vitamin D3 (Cholecalciferol)

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (Cholecalciferol) — an oral solution of vitamin D in a refined olive oil solution

SUMMARY:
This is a three-arm unblinded prospective interventional study of vitamin D supplementation in participants with insufficient vitamin D at three different induction and maintenance dosing regimens (high dose, low frequency; medium dose, medium frequency, and low dose, high frequency). Measurements of serum vitamin D will take place at 4, 8, 12, 24, and 36 weeks, and will be compared to determine which regimen was most effective at achieving and maintaining ideal serum vitamin D levels.

DETAILED DESCRIPTION:
Data obtained from many epidemiological studies suggest that vitamin D deficiency is widespread throughout the world, despite increasing attention to the relationships between vitamin D deficiency and skeletal health as well as many other organ systems. This proposal is designed to optimally replace vitamin D deficient subjects with oral vitamin D solution (Dibase) among a well-characterized population whose mean vitamin D level have been established. In a recent nationwide study, this research team established that the country of Armenia has marginal levels of 25-hydoxyvitamin D among a free-living population of pre- and postmenopausal women: the average level was 19.76 ng/mL with 54% of subjects showing levels that are clearly insufficient. Equally impressive is the finding that fully 20% of women over 65 years of age, have levels that are below 12 ng/mL (< 30 nmol/l).

Following consent, all participants will receive a unique participant identification number, and will then complete a brief questionnaire regarding demographics, selected medical history, and contact information. All participants will then be directed to the EcoSense laboratory, where they will provide blood sample via venipuncture for vitamin D.

For those participants with a 25-hydroxyvitamin D level of less than 30 ng/mL, they will be called back to EcoSense laboratory where they will provide blood sample via venipuncture for calcium, and then brought to the Osteoporosis Center, where they will be randomly allocated into one of three treatment groups.

Participants will be instructed on how to dose the supplement as appropriate for their assigned arm, and then receive 4 weeks of the vitamin D supplement. Participants will return to the Osteoporosis Center at the end of week 4 to obtain an interval history, be assessed for any adverse reactions, compliance, or symptoms of infection or illness. Blood samples will be obtained at weeks 4, 8, 12, 24, and 36 for measurement of 25-hydroxyvitamin D and calcium at the collaborating laboratory as described above, and all participants will be informed of their lab test results as they become available.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75
* Willing to participate in the study
* No vitamin D supplements for at least 1 year

Exclusion Criteria:

* Not meeting inclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Vitamin D level | Baseline, 48 months
  This is to examine the optimal repletion strategy for individuals with hypovitaminosis D. Blood tests will be performed to determine vitamin D levels.
VDBP level | Baseline, 48 months
  This is to examine the optimal repletion strategy for individuals with hypovitaminosis D. Blood tests will be performed to determine Vitamin D Binding Protein (VDBP) levels.

CONTACTS AND LOCATIONS:
Overall Officials: John Bilezikian, MD, Principal Investigator — Professor of Medicine
Locations (1):
- Osteoporosis Center of Armenia, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No